CLINICAL TRIAL: NCT01055236
Title: Hydroxyzine for the Prevention of Pruritus and Nausea Vomiting From Spinal Morphine in Patients Having Transabdominal Hysterectomy Under Combined Spinal-general Anesthesia: A Randomized Control Trial
Brief Title: Hydroxyzine for the Prevention of Pruritus From Spinal Morphine in Transabdominal Hysterectomy Patients
Acronym: TAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Dr. Phuriphong Songarj, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 168/2550(EC1)
Record Dates: First submitted 2010-01-06; First posted 2010-01-25 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2008-12

CONDITIONS: Pruritus; Nausea; Vomiting
Keywords: sedation
MeSH Terms: conditions — Pruritus; Nausea; Vomiting | interventions — Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydroxyzine (Placebo Comparator)
  Interventions: Drug: hydroxyzine
- placebo (Placebo Comparator): starch tablet
  Interventions: Drug: hydroxyzine

INTERVENTIONS:
Drug: hydroxyzine — 75 mg of hydroxyzine orally as premedication drugs at least half an hour before operation.
  Other Names: atarax

SUMMARY:
Hydroxyzine is one of antihistamines that antagonizes H1 receptor, and it's effects are reducing pruritus, nausea/vomiting, and the mild effect of sedation.With these effects Hydroxyzine should be used in the prevention of these symptoms.

DETAILED DESCRIPTION:
80 patients scheduled for elective transabdominal hysterectomy under combined spinal-general anesthesia. they were randomized to receive either hydroxyzine 75 mg and midazolam 7.5 mg (ATR group) or placebo and midazolam 7.5 mg (control group) as premedication at least half an hour before operation. Clinical data (vital signs, pruritic score, nauseous score, sedation score, etc) was recorded at preoperative, intraoperative and 48-hour postoperative periods. All patients had spinal block with 0.5% heavy bupivacaine 2 ml with 0.3 mg preservative free morphine and general anesthesia with thiopental sodium 250-300 mg as induction, intubated with atracurium 0.6 mg/kg and maintenance with nitrous oxide, oxygen and isoflurane. Conventional reversal technique was done in all patients. Fentanyl intravenous was used for pain as needed, chlopheniramine syrup 2 tsp (4mg/10 ml) every 4 hours was used for pruritus and ondansetron intravenous (8 mg) was used for nausea/vomiting in postoperative period. The results were reported in number of patients or percent of patients who were suffered from pruritus, nausea, vomiting or sedation.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification 1-2
* Age from 18-60 years old
* Body mass index (BMI) below 35
* Accepted combined spinal-general anesthesia

Exclusion Criteria:

* Previous history of Hydroxyzine allergy
* Underlying diseases of urticaria, pruritus, nausea vomiting and motion sickness
* Previous complications of procedure or anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
successful treatment of pruritus | 48 hour

SECONDARY OUTCOMES:
successful treatment of nausea or vomiting | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Phuriphong Songarj, MD, Study Director — Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand